CLINICAL TRIAL: NCT02266108
Title: ESTIMA: Economic and Social Empowerment To Increase Upwards Mobility Among Women
Brief Title: Economic and Social Empowerment To Increase Upwards Mobility Among Women
Acronym: ESTIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Elizabeth Reed, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 140523
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Sexually Transmitted Infections; Human Immunodeficiency Virus
Keywords: Sexually Transmitted Infections; Female Sex Workers
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESTIMA intervention (Experimental): This group is randomized to receive the ESTIMA intervention and will be followed for 12 months for follow-up.
  Interventions: Behavioral: ESTIMA Intervention
- Wait-list control (Other): This group will receive standard of care (education as well as referrals to testing and treatment). After 12 months of follow-up, this group will receive the ESTIMA intervention.
  Interventions: Behavioral: ESTIMA Intervention

INTERVENTIONS:
Behavioral: ESTIMA Intervention — This study involves the evaluation of ESTIMA, a microfinance and gender equity intervention among women working as sex workers in Tijuana, Mexico.

SUMMARY:
The proposed research aims to pilot a multi-strategy structural intervention combining community mobilization to promote gender equity alongside an economic intervention (microfinance and business training) in order to reduce gender-based violence and HIV risk among female sex workers (FSW) in Tijuana, Mexico. The program will be called ESTIMA: "Economic and Social Empowerment To Increase Upwards Mobility Among Women." The evaluation will employ a randomized controlled design, recruiting FSW (n=120, 60 in each arm) who will be randomized to: 1) ESTIMA (gender equity/community mobilization program and economic intervention) or 2) a wait-list control group. For this preliminary work, at 12 months follow-up, we hypothesize that compared to control participants, intervention participants will have: 1) significantly greater economic security (e.g. decreased debt, increased income, decreased number of sex trades) and 2) significantly greater perceived collective power (i.e. collective efficacy) to address gendered power imbalances within social structures and the community. The long-term goal of this program, upon future refinement and large scale implementation, is to reduce HIV risk behaviors, STI/HIV, GBV, and ultimately, alleviate a multitude of health burdens among women. Furthermore, we expect that such work will highlight the need for HIV prevention initiatives in Mexico, and elsewhere, to more broadly consider women's 'life contexts' - addressing economic and social burdens in women's lives, to reduce the burden of poverty, gender, and HIV, as well as the intersection of these among women.

DETAILED DESCRIPTION:
The ESTIMA program will consist of the 1) Via microfinance program, which includes providing women with monetary loans as a group (approximately 10 women, with repayment as a group) and training them to initiate a business or other investment endeavor, and 2) gender equity community mobilization, which involves initiating groups of women (i.e. collectives) and engaging in social action within the community, with a focus on addressing issues relevant to gender inequities and women's economic mobility and power (such as client or police violence/harassment). Like the IMAGE program in South Africa, community mobilization will be incorporated into the Via microfinance trainings.

Priorities of mobilization efforts will be identified by the ESTIMA collectives, and facilitated by the election of collective leaders. As part of the microfinance efforts, women will be provided with a loan of up to $200 each and will support each other by agreeing to all be responsible to repay the loan as a group. While the amount is small, women can take out more money with subsequent loans to help them support the business.

The outcome evaluation of ESTIMA will employ a randomized controlled design. From the parent study (Dr. Brouwer, PI;R01 DA028692), we will recruit at least 120 participants in expectation to afford a final sample size of at least 48 in each group (using a conservative estimate of 80% retention). Eligible and willing participants will be randomized to treatment assignment (ESTIMA or wait-list control group) using a randomizer software package, after baseline data collection for the proposed research. The wait-list control group will be provided with referrals to local FSW support organizations, as the standard of care, and will receive ESTIMA subsequent to the 12 month follow-up data collection. ESTIMA will involve groups of approximately 10 women each; groups will initiate once sufficient numbers are enrolled (i.e. groups will be staggered in initiation of the ESTIMA program). Data collection will include a behavioral survey as well as HIV/STI testing.

This combined program addresses economic vulnerability while also supporting women via community mobilization to address challenging social conditions at work, in the community, and at home. This work affords an opportunity to evaluate the efficacy of a microfinance-based initiative to improve health outcomes among an economically vulnerable population of women, many who have been trafficked into sex work, and who face dire economic circumstances to support their families and children. The randomized controlled evaluation design will be among the first implemented among sex workers and among the few implemented globally to evaluate a microfinance-based program in terms of improving health outcomes. Such a robust design will be key to providing evidence needed regarding the efficacy of the ESTIMA program, and implications of the utility of microfinance as a means of HIV prevention among this population.

ELIGIBILITY:
Inclusion Criteria:

* Biologically female,
* At least 18 years old,
* Ability to Speak English or Spanish
* Report having exchanged sex for money, goods, shelter or drugs within the last month,
* Live in Tijuana or its suburbs and have no plans to permanently move over the next 18 months
* Willing and able to provide informed consent
* Agree to receive antibiotic treatment for Chlamydia, gonorrhea and syphilis if they test positive

Exclusion Criteria:

* Not be a part of a recent behavioral intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reed, ScD, Principal Investigator — University of California, San Diego
Locations (1):
- Los Ninos De Baja California, Tijuana, Estado de Baja California, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ESTIMA Intervention | Wait-list Control
Started | 80 | 71
Completed | 80 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ESTIMA Intervention | Wait-list Control | Total
Number analyzed (Participants) | 80 | 71 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 71 | 151
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12) | 37 (11) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 71 | 151
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 2 | 1 | 3
  White | 20 | 23 | 43
  More than one race | 29 | 31 | 60
  Unknown or Not Reported | 28 | 14 | 42
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 80 | 71 | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decreased Economic Vulnerability
Description: Economic vulnerability was measured by asking women about several financial challenges creating urgency in their work. We also measured income.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ESTIMA Intervention | Wait-list Control
Number analyzed (Participants) | 80 | 71
Participants | 51 | 37

2. Primary Outcome: Number of Participants With Increased Collective Efficacy
Description: improved reported support from other women; increased sense of unity within group, increased sense of belonging
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | ESTIMA Intervention | Wait-list Control
Number analyzed (Participants) | 80 | 71
Participants | 42 | 30

3. Primary Outcome: Decreased Sexually Transmitted Infections
Description: decreased reported Sexually Transmitted Infections
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ESTIMA Intervention | Wait-list Control
Number analyzed (Participants) | 80 | 71
Participants | 26 | 30

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | ESTIMA Intervention | Wait-list Control
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/71
Other Adverse Events (participants affected / at risk) | 0/80 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT02266108/Prot_SAP_000.pdf